CLINICAL TRIAL: NCT00001073
Title: A Randomized Phase III Trial of Oral Isotretinoin Versus Observation for Low-Grade Squamous Intraepithelial Lesions in HIV-Infected Women
Brief Title: Safety and Effectiveness of Giving Isotretinoin to HIV-Infected Women to Treat Cervical Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 293; 11269 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Cervix, Dysplasia
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Cervix Dysplasia; Cervix Diseases; Isotretinoin; Cervical Intraepithelial Neoplasia; Cervix Neoplasms; Keratolytic Agents
MeSH Terms: conditions — HIV Infections; Uterine Cervical Dysplasia; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Uterine Cervical Diseases; Uterine Cervical Neoplasms | interventions — Isotretinoin

INTERVENTIONS:
Drug: Isotretinoin

SUMMARY:
The purpose of this study is to see if it is safe and effective to give isotretinoin to HIV-infected women with cervical tumors to prevent these tumors from becoming cancerous.

Cervical tumors are found in both HIV-infected and HIV-negative women. However, HIV-infected women are at a greater risk, and often their tumors become cancerous more quickly than those in HIV-negative women. Isotretinoin may be able to prevent this from happening. However, since these tumors tend to disappear over time, many doctors are hesitant to give their patients isotretinoin since this drug causes birth defects. This study looks at whether it is better to treat cervical tumors in HIV-infected women or to wait and see if they will disappear by themselves.

DETAILED DESCRIPTION:
Cervical neoplasia is frequently seen in HIV-infected women, apparently resulting from immunosuppression and common risk factors, including sexual behavior patterns. In HIV seronegative women, progression of preinvasive neoplasia is relatively slow, and up to 40 percent of low grade squamous intraepithelial lesions (grade I CIN/HPV-associated changes) regress to a normal appearance over time. Many clinicians have opted not to treat CIN I/HPV-associated changes due to this high spontaneous regression rate. Currently, retinoids, principally isotretinoin, are the most consistently effective medical therapy for CIN/HPV-associated changes, but use of isotretinoin in HIV-infected patients has not been extensively documented. (AS PER AMENDMENT 6/10/97)

Patients are randomized to receive oral isotretinoin for 6 months or be observed only for 6 months, with 12 additional months of follow-up. [AS PER AMENDMENT 7/23/99: Follow-up time has been decreased to 9 months from the last patient enrolled.]

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are an HIV-positive female.
* Are at least 13 years old. (Need consent of parent or guardian if under 18.)
* Have cervical tumors, as determined by a biopsy performed by a doctor.
* Agree to use both condoms and the pill during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have received certain cancer therapies (such as chemotherapy) within the past 3 or 4 months.
* Have had a hysterectomy (uterus removed) within the past 4 months.
* Are taking tetracycline or Vitamin A.
* Have taken certain medications. (Approved anti-HIV drugs and medications to prevent AIDS-related opportunistic infections are okay.)
* Are pregnant.

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Robinson, Study Chair; Mitchell Maiman, Study Chair
Locations (40):
- United States (37):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - USC CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Usc La Nichd Crs, Los Angeles, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - San Mateo County AIDS Program, San Mateo, California
  - Howard University Hosp., Div. of Infectious Diseases, ACTU, Washington D.C., District of Columbia
  - South Florida CDC Ft Lauderdale NICHD CRS, Fort Lauderdale, Florida
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Univ. of Chicago - Dept. of Peds., Div. of Infectious Disease, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Tulane Med. Ctr. - Charity Hosp. of New Orleans, ACTU, New Orleans, Louisiana
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Bmc Actg Crs, Boston, Massachusetts
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - Univ. of Nebraska Med. Ctr., Durham Outpatient Ctr., Omaha, Nebraska
  - NJ Med. School CRS, Newark, New Jersey
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Memorial Sloan-Kettering Cancer Ctr., New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington
  - UW School of Medicine - CHRMC, Seattle, Washington
- Puerto Rico (2):
  - Puerto Rico-AIDS CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan
- Mbeya Med. Research Program, Mbeya Referral Hosp. CRS, Mbeya, Tanzania

REFERENCES:
- [Background] Robinson WR, Morris CB. Cervical neoplasia. Pathogenesis, diagnosis, and management. Hematol Oncol Clin North Am. 1996 Oct;10(5):1163-76. doi: 10.1016/s0889-8588(05)70391-9. PMID 8880203